CLINICAL TRIAL: NCT01932099
Title: The Direct Flow Medical TranScatheter Aortic Valve RepLacement System US Feasibility Trial
Brief Title: TranScatheter Aortic Valve RepLacement System US Feasibility Trial
Acronym: SALUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Direct Flow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP 011; G120160 (Other: Direct Flow Medical, Inc.)
Record Dates: First submitted 2013-08-20; First posted 2013-08-30 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Aortic Valve Stenosis
Keywords: pathological constriction; restricted outflow, stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Constriction, Pathologic | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm feasibility study (Experimental): Prospective, multi-center, single arm feasibility study. Subjects will include patients with severe aortic valve stenosis who require replacement of their native aortic valve. The intervention is transcatheter aortic valve replacement.
  Interventions: Device: Transcatheter aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Direct Flow Medical Transcatheter Aortic Valve System is indicated for use in aortic stenosis for patients at extreme surgical risk for aortic valve replacement.
  Other Names: Direct Flow Medical aortic valve system; TAVR

SUMMARY:
A study to assess the safety and effectiveness of the Direct Flow Medical aortic valve system. This is for people with severe aortic stenosis who are not well enough to undergo a surgical repair. The delivery of this device is done via the femoral artery.

DETAILED DESCRIPTION:
The Direct Flow Medical Transcatheter Aortic Valve System is indicated for symptomatic patients who require replacement of their native aortic valve and have a predicted operative mortality or serious morbidity risk of equal or greater 50% at 30 days with surgical aortic valve replacement or are deemed unsuitable for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has severe senile degenerative aortic valve stenosis determined by resting or dobutamine stress echocardiogram and Doppler, or simultaneous pressure recordings at cardiac catheterization defined as: mean gradient >40 mmHg or peak jet velocity >4.0 m/s and an aortic valve area ≤0.8 cm2 or aortic valve area index ≤0.5 cm2/m2.
2. The patient has moderate to severe symptoms from aortic valve stenosis (NYHA Functional Class ≥III).
3. The patient must have a predicted risk of operative mortality or serious irreversible morbidity of >50% at 30 days, or be deemed not suitable for surgery for other reasons. This conclusion shall be based on consensus of one cardiologist and two cardiac surgeons at the investigational site after careful consideration of the patient's STS risk score and co-morbidities, and after at least one of the surgeons participating in the decision has personally examined the patient.
4. The patient been informed of the nature of the study, agrees to its provisions, is willing to comply with protocol-specified follow-up evaluations and has provided written informed consent, approved by the appropriate IRB.

Exclusion Criteria

1. Left ventricular ejection fraction (LVEF) <20% determined by resting echocardiogram
2. Patients with an acute MI within 30 days preceding the index procedure.
3. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the study procedure
4. Patients with impaired renal function (estimated Glomerular Filtration Rate [eGFR] <20cc/min, calculated from serum creatinine by the Cockcroft-Gault formula)
5. Patients with a platelet count of <50,000 cells/mm³ or a WBC < 1000 cells/mm³ within 7 days prior to index procedure.
6. Patients with a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, or who will refuse transfusion.
7. Patients who have received any organ transplant or are on a waiting list for any organ transplant.
8. Patients with known other medical illness (e.g. carcinomas, chronic liver disease, chronic renal disease or chronic end stage pulmonary disease) or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation or is associated with a life expectancy of less than one year, or expectation that patient will not improve despite treatment of aortic stenosis.
9. Patients with known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, and/or contrast sensitivity that cannot be adequately pre-medicated.
10. Patients with a history of a stroke or transient ischemic attack (TIA) within the prior 6 months.
11. Patients with an active gastrointestinal (GI) bleeding within the prior 6 months.
12. Patients presenting with hemodynamic instability or cardiogenic shock defined by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
13. Patients who have a planned treatment with any other investigational device or procedure during the study period, or who are currently participating in an investigational drug or another device trial
14. Any planned surgical, percutaneous coronary or peripheral procedure to be performed prior to the 30 day follow-up from the TAVR procedure.
15. Untreated clinically significant coronary artery disease requiring revascularization
16. Trans-esophageal echocardiography (TEE) is contraindicated
17. Active endocarditis or sepsis within 6 months prior to the study procedure
18. Dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)
19. Congenital bicuspid or unicuspid valve determined by echocardiography
20. Prior aortic or mitral valve surgery or pre-existing prosthetic heart valve in any position
21. Native valve annulus diameter is <19mm or >26mm determined by the screening CT scan
22. Extreme asymmetrical calcification of the native aortic valve determined by the screening CT scan
23. Echocardiographic evidence of intra-cardiac mass, thrombus, vegetation, or spontaneous echo contrast in the left atrium
24. >3+ aortic regurgitation, mitral regurgitation or tricuspid regurgitation
25. Moderate to severe mitral stenosis
26. Thoracic aortic aneurysm (TAA) or abdominal aortic aneurysm (AAA) >5.0 cm
27. Presence of an endovascular stent graft for treatment of AAA or TAA 28 Hypertrophic obstructive cardiomyopathy

29. Patients with severe peripheral arterial disease that precludes sheath vascular access (e.g. luminal diameter less than 6.5 mm, severe obstructive calcification or severe tortuosity)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from all cause mortality/Device success | 6 months post procedure
  Absence of procedural mortality AND correct positioning of a single prosthetic heart valve into the proper anatomic location AND Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient less than 20 mmHg or peak velocity less than 3m/s, AND no moderate or severe prosthetic valve regurgitation.

SECONDARY OUTCOMES:
Early Safety | 30 Days
  Early Safety: as a composite of
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute Kidney Injury - Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complications
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVR, or SAVR)
Clinical Efficacy | 6 months,and annually at 1 to 5 years
  Clinical Efficacy will be evaluated as a composite of:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Hospitalization for valve-related symptoms or worsening congestive heart failure† (including reporting of days hospitalized)
  * NYHA Class III or IV
  * Prosthetic heart valve dysfunction (mean aortic valve gradient ≥20 mm Hg, EOA ≤0.9-1.1 cm2‡ and/or DVI <0.35, AND/OR moderate or severe prosthetic valve regurgitation*)
Time-related Valve Safety | 30 days, 6 months and annually at 1 to 5 years
  Time-related valve safety will be evaluated as a composite of:
  * Structural valve deterioration:
    * Valve-related dysfunction (mean aortic valve gradient (mean aortic valve gradient ≥20 mm Hg, EOA ≤0.9-1.1 cm2[Depending on body surface area] and/or DVI <0.35, AND/OR moderate or severe prosthetic valve regurgitation [VARC defined])
    * Requiring repeat procedure (TAVR or SAVR)
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thromboembolic events (e.g., stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy (e.g., trauma)
Clinical Endpoints | 30 days, 6 months and annually at 1 to 5 years.
  Individual Endpoints
  * All-cause mortality
  * Cardiovascular mortality
  * Non-cardiovascular mortality Myocardial Infarction
  * Peri-procedural MI (<72 hours after the index procedure)
  * Spontaneous MI (>72 hours after the index procedure) Neurological Events
  * Stroke
    * Ischemic stroke
    * Hemorrhagic stroke
    * Undetermined
  * Disabling Stroke
  * Non-disabling stroke
  * Transient ischemic attack Bleeding Complications
  * Life-threatening or disabling bleeding
  * Major bleeding
  * Minor bleeding Acute Kidney Injury (AKIN Classification)
  * Stage 1 acute kidney injury
  * Stage 2 acute kidney injury
  * Stage 3 acute kidney injury Vascular Complications
  * Major vascular complications
  * Minor vascular complications
  * Percutaneous closure device failure Prosthetic Valve Dysfunction
  * Prosthetic Aortic Valve Stenosis
  * Prosthesis-Patient Mismatch
  * Prosthetic Aortic Valve Regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: E. Murat Tuzcu, MD, Principal Investigator — The Cleveland Clinic; Patrick M McCarthy, MD, Principal Investigator — Northwestern Memorial Hospital
Locations (6):
- United States (6):
  - UC Davis Medical Center, Sacramento, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University Hospital, St Louis, Missouri
  - Columbia Univ. Medical Center, New York, New York
  - Cleveland CLinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided